CLINICAL TRIAL: NCT01857024
Title: Renvela® Post-Marketing Observational Study to Monitor the Clinical Use in Adult Hyperphosphataemic Chronic Kidney Disease Patients Not On Dialysis With Serum Phosphorus ≥1.78 mmol/L
Brief Title: Post Authorisation Safety Study of Renvela® in Chronic Kidney Disease Patients Not on Dialysis With Hyperphosphataemia
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: SVCARB06009
Record Dates: First submitted 2013-05-13; First posted 2013-05-20 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Hyperphosphataemia; Chronic Kidney Disease
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic | interventions — Sevelamer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sevelamer carbonate (Renvela®) — 800 mg tablets or 2.4 g powder for oral suspension should be administered as instructed in the Renvela® SmPC.

SUMMARY:
The primary objective of this study is to assess in a post-approval clinical setting the safety profile of sevelamer carbonate (Renvela®) tablets and powder in adult hyperphosphataemic chronic kidney disease (CKD) patients not on dialysis with serum phosphorus ≥1.78 mmol/L. Patients will be treated in accordance with the Renvela® Summary of Product Characteristics (SmPC) and followed according to the investigator's standard clinical practice management. Each patient will be followed up for 12 months or up to the time they start dialysis, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chronic Kidney Disease (CKD) patients not on dialysis with serum phosphorus ≥ 1.78 mmol/L.
* Prescribed Renvela (800 mg tablets or 2.4 g powder for oral suspension) in accordance with the Renvela SmPC.
* Provide signed informed consent (patient or their legally authorised representative)

Exclusion Criteria:

* N/A

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Chronic Kidney Disease (CKD) patients not on dialysis with serum phosphorus ≥ 1.78 mmol/L.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Frequency of non-serious and Serious Adverse Drug Reaction (ADRs) | 12 Months
  Assess safety profile of Renvela tablets and powder

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (26):
- Austria (2):
  - Graz
  - Linz
- Aalborg, Denmark
- France (5):
  - Cabestany
  - Dijon
  - Lille
  - Saint-Laurent-du-Var
  - Toulouse
- Germany (5):
  - Berlin
  - Dortmund
  - Hanover
  - Mettmann
  - Wiesbaden
- Italy (7):
  - Acireale
  - Milan
  - Naples
  - Palermo
  - Pavia
  - Pesaro
  - Rome
- Netherlands (4):
  - Amsterdam
  - Breda
  - Dordrecht
  - Leiden
- Spain (2):
  - Madrid
  - Valencia